CLINICAL TRIAL: NCT01080339
Title: Change in Cardiometabolic Risk Factors During an Interactive Fitness Program: An Exploratory Sub-study
Brief Title: Substudy of Change in Cardiometabolic Disease (CMD) Risk Factors During an Interactive Fitness Program
Acronym: EXCEL
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit participants.
Sponsor: Boston Children's Hospital (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sarah de Ferranti, MD, Children's Hospital Boston
Other Study IDs: 09-12-0611
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Insulin Resistance
Keywords: insulin resistance; cardiovascular risk; physical activity; child
MeSH Terms: conditions — Insulin Resistance; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Physical Activity and Nutrition: Supervised physical activity in the form of novel gaming and exercise equipment several times per week for 12 weeks will be provided in addition to weekly nutrition education sessions.
- Nutrition Education Only: Children in this group will receive weekly group nutrition sessions, identical to those provided for the Physical Activity + Nutrition group

SUMMARY:
Substudy examining cardiovascular and metabolic risk factor change in children at high risk for future atherosclerosis who are enrolled in a pilot intervention using novel gaming and exercise activities to increase physical activity.

DETAILED DESCRIPTION:
Childhood obesity is increasingly common and is predictive of adult type 2 diabetes and cardiovascular disease (CVD). Recent pediatric studies suggest exercise reduces cardiometabolic risk factors. Despite evidence of its benefits, exercise training prescribed by pediatricians is traditionally vague, developmentally inappropriate, and/or fraught with psychological, financial and practical barriers. There has been recent interest in the use of interactive technologies, also termed "exer-gaming" as a way to translate known positive benefits of exercise into increased physical activity in youth. Initial adult studies demonstrate benefits, yet there are few studies of exer-gaming involving children at increased CVD risk. This project involves a partnership between Children's Hospital Boston and the GoKids Boston Youth Fitness Research and Training Center at UMass Boston, featuring an interdisciplinary team of researchers and clinicians from pediatric cardiology, prevention, nursing, exercise physiology, and behavior change. Participants are eligible for this substudy based on enrollment in a pilot project evaluating the effects of a state-of-the-art exercise training facility incorporating the latest technology-based exercise games ("exer-games") in Boston Public School elementary children. Effects on CVD risk factor levels including lipids, blood pressure, body composition vascular reactivity, insulin resistance pre and post intervention will be compared to an Advice-Only condition and correlated with activity level. Eligible participants will be identified as part of the baseline measurements of that study and will be offered the chance to participate in the CHB Sub-Study, a two visit observational design.

ELIGIBILITY:
Inclusion Criteria:

* Participation in main intervention study

Exclusion Criteria:

* Unwillingness to comply with study requirements including two visits and data collection procedures

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children attending 3rd-5th grades at select Boston Public Schools will be eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity (HOMA-IR) | 12 weeks
  Homeostasis model assessment of insulin resistance (HOMA-IR) will be measured at baseline and after 12 weeks of physical activity plus nutrition advice intevention, or nutrition-only advice.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D de Ferranti, MD MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Levenson AE, Milliren CE, Biddinger SB, Ebbeling CB, Feldman HA, Ludwig DS, de Ferranti SD. Calorically restricted diets decrease PCSK9 in overweight adolescents. Nutr Metab Cardiovasc Dis. 2017 Apr;27(4):342-349. doi: 10.1016/j.numecd.2016.12.010. Epub 2017 Jan 3. PMID 28228332
- [Derived] de Ferranti SD, Milliren CE, Denhoff ER, Quinn N, Osganian SK, Feldman HA, Ebbeling CB, Ludwig DS. Providing food to treat adolescents at risk for cardiovascular disease. Obesity (Silver Spring). 2015 Oct;23(10):2109-17. doi: 10.1002/oby.21246. Epub 2015 Sep 4. PMID 26337820